CLINICAL TRIAL: NCT03038581
Title: Comparison of Self-inflicted Deep Wrist Injuries to Traumatic Deep Wrist Injuries
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Kisch, MD, University Hospital Schleswig-Holstein
Other Study IDs: 13-054; U1111-1176-0115 (Other: WHO)
Record Dates: First submitted 2015-10-29; First posted 2017-01-31 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Deep Wound; Wrist Injuries
Keywords: Deep wrist injury; Self inflicted; Traumatic wrist injury
MeSH Terms: conditions — Wrist Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Self-inflicted wrist injury: Wrist injury by self-infliction
- Traumatic wrist injury: Wrist injury by not self-inflicted trauma

SUMMARY:
Self-inflicted wrist injuries require special psychiatric knowledge and tactical skills. There is no protocol for treating such injuries. We analyze self-inflicted wrist injuries and compare them to traumatic wrist injuries.

DETAILED DESCRIPTION:
Self-inflicted wrist injuries are regularly treated in hand surgery centers. These injuries involve risks that require special psychiatric knowledge and tactical skills. There is no protocol for treating such injuries. Therefore, the investigators analyze self-inflicted wrist injuries and compare them to traumatic wrist injuries.

ELIGIBILITY:
Inclusion Criteria:

* Deep wrist injury from 2008-2018
* Treated in University Hospital Schleswig-Holstein
* Agreed to retrospective analysis, questionnaires and hand function assessment

Exclusion Criteria:

* Non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with deep wrist injuries that were treated 2008-2018 in University Hospital Schleswig-Holstein
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Hand function | Up to 10 years
  Assessment of hand function by measuring sensibility (2-point-discrimination) and motoric (degree joints)

SECONDARY OUTCOMES:
Psychiatric history | Up to 10 years
  Assessment of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Principal Investigator — University of Schleswig-Holstein, Campus Lübeck, Germany
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No